CLINICAL TRIAL: NCT05286190
Title: Effects Of Ultrasound Guided Caudal Epidural And Transversus Abdominis Plane Block On Postoperative Analgesia In Pediatric Inguinal Hernia Repair Surgeries
Brief Title: Caudal Block and Transversus Abdominis Plane Block in Pediatric Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associate Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017/1123
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Regional Anesthesia; Postoperative Pain, Acute
Keywords: US guided Caudal Epidural Block; US guided Transversus Abdominis Plane Block
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversus Abdominis Plane Block (Active Comparator): US-guided Transversus Abdominis Plane Block was applied with 0.5 ml/kg of %25 Bupivacaine at each side before the surgical incision
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution
- Caudal Epidural Block (Active Comparator): US-guided Caudal Block was applied with 0.7ml/kg of %25 Bupivacaine before the surgical incision
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution

INTERVENTIONS:
Drug: Bupivacaine 0.25% Injectable Solution — Bupivacaine 0.25% Injectable Solution
  Other Names: Marcaine

SUMMARY:
Pediatric inguinal hernia repair (IHR) candidates experiences ordinarily mild to moderate pain, rarely severe pain in the postoperative period. Caudal epidural block (CEB) and transversus abdominis plane block (TAPB) are two effective postoperative analgesia options. In this randomized study, it is aimed to compare the effects of CEB and TAPB on postoperative pain scores, additional analgesic requirement, postoperative nausea and vomiting incidence, procedural complications, family and surgeon satisfaction, length of hospital stay, chronic pain development in pediatric bilateral open IHR.

DETAILED DESCRIPTION:
Inguinal hernia repair (IHR) is the second common operation in pediatric surgery practice following appendectomy and bilateral repair is needed in 10.9% of the cases due to presence of contralateral inguinal hernia. After IHR, the children generally experiences mild to moderate pain, and occasional severe pain. For pediatric population the prevalence of chronic pain after IHR is 5% which is a solid cause for severe pain.

Adequate pain control is a crucial part of perioperative management to reduce morbidity and ensure family and patient satisfaction especially after pediatric surgeries. Although there are substantial studies to show how to assess and manage the postoperative pain in children, the pain control is often not achieved. Several analgesic regimens including systemic medications and/or regional analgesia methods may be preferred by clinicians. As previous studies revealed; best combination for pain management after pediatric IHR is still obscure.

Caudal epidural block (CEB) and transversus abdominis plane block (TAPB) are the two regional analgesia methods which may be chosen for multimodal analgesia. CEB is accepted as gold standard for lower abdominal surgeries in children which diminishes somatic and visceral pain with a duration of 6 hours. TAPB is another regional analgesia method which covers only somatic pain up to 24 hours postoperatively with lower complication rates compared to CEB. The results of clinical studies examining the effects of CEB and TAPB on early postoperative pain after pediatric IHR are conflicting. Currently, the effects of these blocks on the incidence of chronic pain after pediatric IHR is not well-investigated in the literature. As a matter of fact, there are no recommendations for bilateral IHR in pediatric postoperative pain guidelines, despite these surgical procedures being an independent risk factor for severe pain.

In this randomized study, it is aimed to compare the effects of ultrasound (US) guided CEB and TAPB on postoperative analgesia. Our hypothesis was that bilateral TAPB block will be equally effective as CEB in the early postoperative period and the analgesic duration will be longer than CEB. Our primary outcome was FLACC (face, legs, activity, cry, consolability) scores in postoperative 24 hours. The secondary outcomes included additional analgesic requirements, postoperative nausea vomiting incidence, procedural complications, length of hospital stay, family and surgeon satisfaction and chronic pain development at the postoperative 2nd month.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 1-7 years who were scheduled for elective bilateral open IHR included in the study

Exclusion Criteria:

* Patients with relative or absolute contraindications to TAPB or CEB, patients with chronic constipation or chronic pain disorders that may affect the evaluation of postoperative pain scores, patients who underwent emergency surgery, and patients with a history of allergic reaction to local anesthetics were excluded from the study.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
FLACC SCORES (FACE, LEG, ACTIVITY, CONSOLABILITY, CRY) | Up to 24 hours
  It includes five categories of behavior, each scored on 0-2 point scale so that total score ranges from 0 to 10. Total scores of 0-3 is defined as mild, 4-7 as moderate, and 8-10 as severe pain.

SECONDARY OUTCOMES:
PONV (Postoperative nausea and vomiting) | Up to 24 hours
  Number of patients with nausea vomiting
Additional analgesic requirement | Up to 24 hours
  Number of patients who require paracetamol (15 mg/kg) and tramadol (1 mg/kg)
Family satisfaction | Up to 24 hours
  A 3-point scale (satisfied:3; neutral:2, dissatisfied:1)
Surgeon satisfaction | Up to 24 hours
  A 3-point scale (satisfied:3; neutral:2, dissatisfied:1)
Complications | Up to 24 hours
  Possible complications related to caudal and transversus abdominis plane block (hematoma, infection and perforation)
Revised Bieri faces pain scale | At postoperative 2nd month
  Revised Bieri faces pain scale used for assessment of chronic pain. Score the chosen face 0,2,4,6,8,10 counting left to right so '0'=no pain and '10'=very much pain
Length of hospital stay | Through study completion, an average of 1 week
  Hospitalisation

CONTACTS AND LOCATIONS:
Locations (1):
- Meltem Savran Karadeniz, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Derived] Polat H, Senturk E, Savran Karadeniz M, Bingul ES, Emre Demirel E, Erginel B, Tugrul KM. Effects of ultrasound guided caudal epidural and transversus abdominis plane block on postoperative analgesia in pediatric inguinal hernia repair surgeries. J Pediatr Urol. 2023 Apr;19(2):213.e1-213.e7. doi: 10.1016/j.jpurol.2022.11.005. Epub 2022 Nov 15. PMID 36446689